CLINICAL TRIAL: NCT03993158
Title: Prospective Cohort Study for Newborns From Patients Treated With ART in Clinical Reproductive Medicine Management System/Electronic Medical Record Cohort Database (CCRM/EMRCD)
Brief Title: Newborns From Patients Treated With ART (Assisted Reproductive Technology)
Status: Recruiting | Type: Observational
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Yingpu Sun, Director of Reproductive Medical Center, The First Affiliated Hospital of Zhengzhou University
Other Study IDs: RMCZZU-Birth cohort study
Record Dates: First submitted 2019-06-18; First posted 2019-06-20 (Actual); Last update posted 2019-06-20 (Actual); Status verified 2019-06

CONDITIONS: Health Related

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Prospective Cohort Study for Newborns from patients treated with ART was set up to investigate the short- and long-term health consequences in Reproductive Medical Center, First Affiliated Hospital of Zhengzhou University, China.

DETAILED DESCRIPTION:
Since the last twenty years, thousands of babies were born from infertile couples treated in our center. However, the short, and especially the long term prognosis of these children were barely known.

Since last decade, Clinical Reproductive Medicine Management System/Electronic Medical Record Cohort Database (CCRM/EMRCD) has been used in Reproductive Medical Center, First Affiliated Hospital of Zhengzhou University, and Henan Province Key Laboratory for Reproduction and Genetics. Information of patients (POI, PCOS, Endometriosis, azoospermia, ect) were recorded comprehensively. In addition, information of each newborn from our center has also been kept in CCRM/EMRCD. The current project plans to recruit these newborn babies in our center. Biological samples, questionnaires and short/long term health data will be collected. The study is aimed to provide evidence for Newborns from patients treated with ART prognosis.

ELIGIBILITY:
Inclusion Criteria:

* All newborns from patients treated with ART in our center.

Exclusion Criteria:

-

Max Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All newborns from patients treated with ART in our center.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2010-01-01 (Actual); Primary Completion 2050-12-31 (Estimated); Study Completion 2050-12-31 (Estimated)

PRIMARY OUTCOMES:
Birth weight | At delivery
  Weight of newborns recorded in Kilogram
Number of newborns with Congenital malformations | At delivery
  Any newborns with Congenital malformations will be recorded

SECONDARY OUTCOMES:
Height development of newborns | at age of 1 month, 3 months, 6months, 1 year, 3 years and 6 years
  Record the height changes (in centimeters)

CONTACTS AND LOCATIONS:
Locations (1):
- Reproductive Medical Center, First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China

REFERENCES:
- [Background] Giorgione V, Parazzini F, Fesslova V, Cipriani S, Candiani M, Inversetti A, Sigismondi C, Tiberio F, Cavoretto P. Congenital heart defects in IVF/ICSI pregnancy: systematic review and meta-analysis. Ultrasound Obstet Gynecol. 2018 Jan;51(1):33-42. doi: 10.1002/uog.18932. PMID 29164811
- [Background] Wagenaar K, Huisman J, Cohen-Kettenis PT, Delemarre-van de Waal HA. An overview of studies on early development, cognition, and psychosocial well-being in children born after in vitro fertilization. J Dev Behav Pediatr. 2008 Jun;29(3):219-30. doi: 10.1097/DBP.0b013e318173a575. PMID 18550992